CLINICAL TRIAL: NCT04082195
Title: Impact of Digital Health Education Intervention - Fooya on Health Awareness Around Eating Right and Physical Activity of School Going Children in Chennai
Brief Title: Impact of A Mobile Game on Pediatric Nutrition and Physical Activity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Center for Communication and Change India (Other)
Collaborators: Johns Hopkins University (Other); Carnegie Mellon University (Other); Hofstra University (Other); FriendsLearn Inc. (Unknown); The Mithra Trust (Unknown); Mind in Motion (Unknown); Seethapathy Clinic & Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00006230
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Pediatric Nutrition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fooya mobile game (Experimental): An arm that receives a mobile-app-based treatment.
  Interventions: Other: Fooya mobile game
- Uno board game (Active Comparator): An arm that receives a non mobile-app-based treatment.
  Interventions: Other: Uno board game

INTERVENTIONS:
Other: Fooya mobile game — An application that incorporates the science and technology of immersive gaming, neuropsychology and cognitive behavior therapy in a mobile health game to target early childhood nutrition literacy and health promotion in a fun and exciting way.
  Arms: Fooya mobile game
Other: Uno board game — A popular board game which is not a mobile app.
  Arms: Uno board game

SUMMARY:
Overweight and obesity in children is on the rise globally and is rapidly growing in urban India. Studies have revealed that obesity is on the rise among children in India with many of them suffering from the problem even before they reach adolescence.

As many as 30 million Indians are overweight, and obesity continues to rise. The National Family Health Survey (NFHS) found that 20% of school children are overweight. NFHS is a large-scale, multi-round survey conducted in a representative sample of households throughout India. The findings from the survey indicate that the prevalence of obesity is increasing in India along with the epidemic proportions worldwide especially in developed countries.

Overweight or obesity is the leading cause of type 2 diabetes, gestational diabetes, hypertension, osteoarthritis, various types of cancers in women like breast cancer and uterine cancer, menstrual disorder and infertility and many more diseases.

To decrease prevalence you have to decrease incidence. More and more young people are at risk of developing diseases like diabetes and if the number of children living with these diseases has to come down, focus has to be on addressing the risk factors and moving the population to a healthier lifestyle through health education/ communication and motivation. To design appropriate interventions for behaviour formation and change, we need to learn more about the underlying factors affecting these unhealthy behaviours.

This study was conducted by the Center for Communication and Change - India, in partnership with the Johns Hopkins Bloomberg School of Public Health Center for Communication Programs, and FriendsLearn (California).

Study Purpose

The specific aim of this research study is to assess the awareness levels among urban, Indian children, with respect to diet and lifestyle behaviours, while also evaluating the influence of a digital health education intervention - fooya!™ among school-age children in India. Specifically, the study objectives will be:

1. Quantify the effectiveness of a digital health education intervention- fooya (an application) on health awareness around eating right and physical activity
2. Find out the current diet and physical activity among urban, children in India and the factors that affect them
3. Assess the extent of their awareness about eating right and physical activity

ELIGIBILITY:
Inclusion Criteria:

* class (grade) 5 students

Exclusion Criteria:

* none

Ages: 10 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2016-12-09 (Actual)

PRIMARY OUTCOMES:
Actual food choice | Immediately after the intervention
  The children were offered a selection of food items to choose from, and the actual selection were documented.

SECONDARY OUTCOMES:
Subjective food choice | Immediately after the intervention
  The children completed surveys to indicate their preferred food items among a list
Knowledge of healthy eating | Immediately after the intervention
  The children completed surveys to indicate their knowledge of healthy eating practice
Knowledge of physical activity | Immediately after the intervention
  The children completed surveys to indicate their knowledge of physical activity

REFERENCES:
- [Derived] Kato-Lin YC, Kumar UB, Sri Prakash B, Prakash B, Varadan V, Agnihotri S, Subramanyam N, Krishnatray P, Padman R. Impact of Pediatric Mobile Game Play on Healthy Eating Behavior: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Nov 18;8(11):e15717. doi: 10.2196/15717. PMID 33206054